CLINICAL TRIAL: NCT02549768
Title: Effect of Dexmedetomidine as Anesthetic Coadjuvant on Plasmatic Cortisol Response in Transsphenoidal Surgery for Pituitary Tumors
Brief Title: Effect of Dexmedetomidine on Plasmatic Cortisol Response in Transsphenoidal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-095
Record Dates: First submitted 2015-09-06; First posted 2015-09-15 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Pituitary Neoplasms
Keywords: Dexmedetomidine; Pituitary; Transsphenoidal; Cortisol
MeSH Terms: conditions — Pituitary Neoplasms; Pituitary Diseases | interventions — Dexmedetomidine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Use of dexmedetomidine during surgery (1 mcg/kg in 10 minutes, then infusion at 0.7 mcg/kg/h)
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Use of crystalloid solution (sodium chloride 0.9%), injection pump programmed with drug "Dexmedetomidine" with 1 mcg/kg in 10 minutes, infusion 0.7 mcg/kg/h.
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Dexmedetomidine — At start of anesthesia, bolus of 1 mcg/kg of dexmedetomidine over 10 minutes and then infusion of 0.7 mcg/kg/h during surgery will be administered.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Sodium Chloride 0.9% — Sodium chloride 0.9% with a pump programmed in same way as Dexmedetomidine pump
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
Use of dexmedetomidine in pituitary tumor resection surgery as adjuvant drug and its relation to cortisol levels during postoperative period.

DETAILED DESCRIPTION:
Transsphenoidal resection of pituitary tumors is the neurosurgical procedure of choice to remove most of the tumors of the sellar region. Sometimes the intervention produces dysfunction of the hypothalamic-pituitary axis, and although most are transient, the risk associated with post-operative hypocortisolism determines its evaluation early in the postoperative period and the possibility of steroidal supplementation posteriorly. It is described that dexmedetomidine can be used as an adjuvant drug in this type of surgery being useful in reduction of total consumption of opioids and anesthetic gases, maintain hemodynamic stability and less time to recovery from anesthesia. Due to its sympatholytic effect, dexmedetomidine has been found to alter the intraoperative common neuroendocrine response generating lower levels of cortisol in the postoperative period than patients in which is not used.

The main objective of this study is to evaluate corticosteroid axis response (cortisol and adrenocorticotropic hormone) in patients undergoing transsphenoidal surgery under anesthesia with dexmedetomidine. A single-center randomized double-blind clinical trial will be conducted that will compare two groups of patients, one of which will be given dexmedetomidine (Dex group) and another group who will receive a placebo (control group). In addition the incidence of perioperative complications (nausea, vomiting, diabetes insipidus), intraoperative hemodynamics and patient comfort. The investigators expect that the normal stress response to surgery measured by cortisol and adrenocorticotropic hormone in the postoperative period will be reduced in the dexmedetomidine arm. This effect should be transient and attributed to use of dexmedetomidine and not to surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II.
* Pituitary tumour: non-functional macroadenoma, Rathke's cleft cyst, acromegaly.
* Normal hypothalamic-pituitary-adrenal axis by hormone levels measurement previous to surgery.

Exclusion Criteria:

* Cushing disease.
* Pituitary apoplexy.
* Craniopharyngioma.
* Chronic corticosteroid use.
* Hemodynamic instability.
* Altered consciousness (Glasgow Coma Scale score less than 15).
* Atrioventricular block in any degree.
* Preoperative bradycardia.
* Alpha 2 agonist use (clonidine, alpha-methyldopa)
* Pregnancy or breast feeding.
* Known allergy to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Cortisol plasmatic levels | 24 hours after surgery
  Venous blood sample

SECONDARY OUTCOMES:
Adrenocorticotropin hormone | One hour after surgery, 24 hours after surgery, 48 hours after surgery
  Venous blood sample
Hemodynamics | From start of anesthesia to end of anesthesia
  Heart rate and arterial pressure
Nausea and vomiting | 24 hours after surgery
  Semiquantitative measure
Pain | 24 hours after surgery
  By visual analogue scale
Patient comfort | 24 hours after discharge from hospital
  Scale ranging from 1 (very unsatisfied) to 5 (very satisfied)
Diabetes insipidus incidence | 24 hours after surgery and 3 months after surgery
  Clinical diagnosis by urine output (polyuria over 3 liters or urine per day) and/or hypernatremia (plasmatic sodium over 145 meq/L)
Cerebrospinal fluid fistula | 3 months after surgery
  Clinical diagnosis made by neurosurgeon
Cortisol plasmatic levels | 1 hour after surgery, 48 hours after surgery, 3 months after surgery
  Venous blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Pedemonte, MD, Principal Investigator — Physician; Pablo Villanueva, MD, Principal Investigator — Assisstant adjunct professor
Locations (1):
- Division de Anestesia - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carrasco CA, Villanueva G P. [Selective use of glucocorticoids during the perioperative period of transsphenoidal surgery for pituitary tumors]. Rev Med Chil. 2014 Sep;142(9):1113-9. doi: 10.4067/S0034-98872014000900004. Spanish. PMID 25517050
- [Background] Hout WM, Arafah BM, Salazar R, Selman W. Evaluation of the hypothalamic-pituitary-adrenal axis immediately after pituitary adenomectomy: is perioperative steroid therapy necessary? J Clin Endocrinol Metab. 1988 Jun;66(6):1208-12. doi: 10.1210/jcem-66-6-1208. PMID 3372683
- [Background] Ali Z, Prabhakar H, Bithal PK, Dash HH. Bispectral index-guided administration of anesthesia for transsphenoidal resection of pituitary tumors: a comparison of 3 anesthetic techniques. J Neurosurg Anesthesiol. 2009 Jan;21(1):10-5. doi: 10.1097/ANA.0b013e3181855732. PMID 19098618
- [Background] Bhana N, Goa KL, McClellan KJ. Dexmedetomidine. Drugs. 2000 Feb;59(2):263-8; discussion 269-70. doi: 10.2165/00003495-200059020-00012. PMID 10730549
- [Background] Gopalakrishna KN, Dash PK, Chatterjee N, Easwer HV, Ganesamoorthi A. Dexmedetomidine as an Anesthetic Adjuvant in Patients Undergoing Transsphenoidal Resection of Pituitary Tumor. J Neurosurg Anesthesiol. 2015 Jul;27(3):209-15. doi: 10.1097/ANA.0000000000000144. PMID 25493927
- [Background] Raekallio MR, Kuusela EK, Lehtinen ME, Tykkylainen MK, Huttunen P, Westerholm FC. Effects of exercise-induced stress and dexamethasone on plasma hormone and glucose concentrations and sedation in dogs treated with dexmedetomidine. Am J Vet Res. 2005 Feb;66(2):260-5. doi: 10.2460/ajvr.2005.66.260. PMID 15757125
- [Background] Mukhtar AM, Obayah EM, Hassona AM. The use of dexmedetomidine in pediatric cardiac surgery. Anesth Analg. 2006 Jul;103(1):52-6, table of contents. doi: 10.1213/01.ane.0000217204.92904.76. PMID 16790625
- [Background] Nomikos P, Ladar C, Fahlbusch R, Buchfelder M. Impact of primary surgery on pituitary function in patients with non-functioning pituitary adenomas -- a study on 721 patients. Acta Neurochir (Wien). 2004 Jan;146(1):27-35. doi: 10.1007/s00701-003-0174-3. Epub 2004 Jan 7. PMID 14740262
- [Background] Bekker A, Haile M, Kline R, Didehvar S, Babu R, Martiniuk F, Urban M. The effect of intraoperative infusion of dexmedetomidine on the quality of recovery after major spinal surgery. J Neurosurg Anesthesiol. 2013 Jan;25(1):16-24. doi: 10.1097/ANA.0b013e31826318af. PMID 22824921